CLINICAL TRIAL: NCT01057173
Title: Transcatheter Versus Surgical Aortic Valve Implantation in Patients With Severe Aortic Valve Stenosis
Brief Title: The Nordic Aortic Valve Intervention Trial
Acronym: NOTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Sahlgrenska University Hospital (Other); Danish Heart Foundation (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Hans Gustav Hørsted Thyregod, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HA2009046
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Critical Aortic Stenosis
Keywords: Heart Valve Disease; Heart Valve Prosthesis; Heart Valve Prosthesis Implantation; Randomized Controlled Trial
MeSH Terms: conditions — Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcatheter Aortic Valve Implantation (Experimental)
  Interventions: Procedure: Transcatheter Aortic Valve Implantation
- Surgical Aortic Valve Replacement (Active Comparator)
  Interventions: Procedure: Surgical Aortic Valve Replacement

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation — Retrograde trans-femoral or trans-subclavian aortic valve implantation with the Medtronic CoreValve System(TM) bio-prosthesis (third generation system, 18 Fr, CE mark approved)
  Other Names: TAVI
  Arms: Transcatheter Aortic Valve Implantation
Procedure: Surgical Aortic Valve Replacement — Conventional surgical aortic valve replacement with a bio-prosthesis using normothermic cardiopulmonary bypass and cold blood cardioplegia cardiac arrest
  Other Names: SAVR
  Arms: Surgical Aortic Valve Replacement

SUMMARY:
A randomized clinical trial of transcatheter aortic valve implantation (TAVI) versus conventional surgical aortic valve replacement (SAVR) in patients older than 70 years of age suffering from severe aortic valve stenosis.

Study hypothesis: TAVI will reduce post-interventional morbidity and mortality compared to SAVR.

DETAILED DESCRIPTION:
BACKGROUND: Transcatheter aortic valve implantation (TAVI) is a new and rapidly evolving treatment option for patients with severe degenerative aortic valve stenosis. Short- and mid-term results with transcatheter valve prostheses are promising in high-risk surgical patients, but long-term results are lacking. TAVI could potentially be an attractive minimally invasive treatment also for patients with moderate and low surgical risk, but no comparison has been made with the standard surgical treatment for aortic valve stenosis.

AIM: To compare TAVI and surgical aortic valve replacement (SAVR) in patients with severe aortic valve stenosis.

POPULATION: All patients with severe degenerative aortic valve stenosis referred for elective or subacute aortic valve intervention will be screened for study eligibility. To be included subjects must be 70 years or older, anatomical and technical eligible for both interventions, expected to survive more than 1 year after the intervention, and able to provide written informed consent. Study exclusion criteria include isolated aortic valve regurgitation or other significant valve disease, coronary artery disease requiring revascularisation at the time of referral, previous open heart surgery, a myocardial infarction or percutaneous coronary intervention within the last year, a cerebral infarction within the previous 30 days, severe renal -, pulmonary -, or infectious disease, and unstable preoperative condition.

DESIGN: The project is a national multicenter randomized clinical trial. Patients fulfilling all inclusion- and no exclusion criteria will be randomized to either TAVI or SAVR. Randomization will be 1:1 with 140 subjects in each group and stratified according to centre, age (70-74 years vs 75 and older), and coronary co-morbidity not requiring revascularisation (yes vs no). Primary outcome will be assessed by a blinded adjudication committee. Patients screened but not included in the study will be followed yearly. Screening and inclusion will commence in December 2009. Inclusion is expected to last 2 to 3 years, and subjects will be followed for 10 years.

INTERVENTIONS: Subjects randomized to TAVI will undergo percutaneous retrograde trans-femoral or trans-subclavian aortic valve implantation with the Medtronic CoreValve(TM) self-expandable bio-prosthesis. Before implantation a balloon dilatation of the aortic annulus will be performed. Subjects randomized to SAVR will undergo conventional surgical aortic valve replacement with a bio-prosthesis on cardiopulmonary bypass in normothermia with cold cardioplegia cardiac arrest. All interventions will be performed under general anaesthesia, and post-interventional medical and anticoagulation treatment will be uniform.

END POINTS: The primary end point is a combined outcome measure consisting of death from any cause, myocardial infarction, and stroke one year after the intervention. Secondary end points are death from any cause, cardiac death, cardiac -, cerebral -, pulmonary -, and renal complications, prosthesis re-intervention, procedure success and - time, admission lengths, functional class, quality of life, prosthesis and left ventricular structure and function. Follow-up visits will be performed after 30 days, 3, 6 and 12 months, and yearly thereafter for a minimum of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have severe degenerative aortic valve stenosis (echocardiographic criteria: AV effective orifice area (EOA) of < 1 cm2, mean AV gradient of > 40 mmHg, or AV peak systolic velocity of > 4.0 m/s)
* Patients must be symptomatic from the aortic valve stenosis (dyspnoea in NYHA-class II or greater, angina pectoris, or syncope), or asymptomatic but with echocardiographic evidence of left ventricular hypertrophy, decreased left ventricular ejection fraction, or atrial fibrillation)
* Patients must be 70 years or older
* Patients must be technical and anatomical eligible for both interventions (as specified by Medtronic CoreValve(TM) for the TAVI procedure) after a formal consult by a cardiologist and a cardiovascular surgeon
* Patients must be expected to survive more than one year after the intervention
* Patients must be able to provide written informed consent as approved by the regional ethical committee after having received adequate information about the study
* Patients must be able and agree to return to all post-procedural follow-up visits

Exclusion Criteria:

* Isolated aortic valve insufficiency
* Other significant heart valve disease requiring intervention
* Coronary artery co-morbidity requiring revascularisation
* Any previous open heart surgery
* Myocardial infarction or percutaneous coronary intervention within the last year
* Stroke or TIA within the last 30 days
* Renal insufficiency requiring hemodialysis
* Pulmonary insufficiency (FEV1 or diffusion capacity < 40% of expected)
* Active infectious disease requiring antibiotics
* Emergency intervention (within 24 hours after the indication for intervention has been made)
* Unstable pre-interventional condition requiring inotropic support or mechanical heart assistance
* A known hypersensitivity or contraindication to heparin or nitinol
* Currently participating in an investigational drug or another device study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Combined rate of death from any cause, myocardial infarction, and stroke | 1 year
  Outcome measures will be defined as suggested by the Valvular Academic Research Consortium (VARC)

SECONDARY OUTCOMES:
Procedural complications | Within first 30 days
Admission lengths (ICU and interventional center) | Within first 30 days
Combined rate of noncardiac and cardiac death, prosthesis reintervention, cardiac-, cerebral-, renal-, and pulmonary complications | 1 year
Functional status (NYHA-classification) and Quality of Life (SF-36) | 1 year
Echocardiographic prosthesis and ventricular structural and functional status | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hans GH Thyregod, MD, PhD, Principal Investigator — Dep. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen University Hospital; Lars Søndergaard, MD, DMSc, Principal Investigator — Dep. of Cardiology, Rigshospitalet, Copenhagen University Hospital
Locations (3):
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen
  - Odense University Hospital, Odense
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Thyregod HG, Sondergaard L, Ihlemann N, Franzen O, Andersen LW, Hansen PB, Olsen PS, Nissen H, Winkel P, Gluud C, Steinbruchel DA. The Nordic aortic valve intervention (NOTION) trial comparing transcatheter versus surgical valve implantation: study protocol for a randomised controlled trial. Trials. 2013 Jan 9;14:11. doi: 10.1186/1745-6215-14-11. PMID 23302232
- [Result] Thyregod HG, Steinbruchel DA, Ihlemann N, Nissen H, Kjeldsen BJ, Petursson P, Chang Y, Franzen OW, Engstrom T, Clemmensen P, Hansen PB, Andersen LW, Olsen PS, Sondergaard L. Transcatheter Versus Surgical Aortic Valve Replacement in Patients With Severe Aortic Valve Stenosis: 1-Year Results From the All-Comers NOTION Randomized Clinical Trial. J Am Coll Cardiol. 2015 May 26;65(20):2184-94. doi: 10.1016/j.jacc.2015.03.014. Epub 2015 Mar 15. PMID 25787196
- [Result] Thyregod HG, Steinbruchel DA, Ihlemann N, Ngo TA, Nissen H, Kjeldsen BJ, Chang Y, Hansen PB, Olsen PS, Sondergaard L. No clinical effect of prosthesis-patient mismatch after transcatheter versus surgical aortic valve replacement in intermediate- and low-risk patients with severe aortic valve stenosis at mid-term follow-up: an analysis from the NOTION trial. Eur J Cardiothorac Surg. 2016 Oct;50(4):721-728. doi: 10.1093/ejcts/ezw095. Epub 2016 Mar 22. PMID 27005980
- [Result] Sondergaard L, Steinbruchel DA, Ihlemann N, Nissen H, Kjeldsen BJ, Petursson P, Ngo AT, Olsen NT, Chang Y, Franzen OW, Engstrom T, Clemmensen P, Olsen PS, Thyregod HG. Two-Year Outcomes in Patients With Severe Aortic Valve Stenosis Randomized to Transcatheter Versus Surgical Aortic Valve Replacement: The All-Comers Nordic Aortic Valve Intervention Randomized Clinical Trial. Circ Cardiovasc Interv. 2016 Jun;9(6):e003665. doi: 10.1161/CIRCINTERVENTIONS.115.003665. PMID 27296202
- [Result] Ngo A, Hassager C, Thyregod HGH, Sondergaard L, Olsen PS, Steinbruchel D, Hansen PB, Kjaergaard J, Winther-Jensen M, Ihlemann N. Differences in left ventricular remodelling in patients with aortic stenosis treated with transcatheter aortic valve replacement with corevalve prostheses compared to surgery with porcine or bovine biological prostheses. Eur Heart J Cardiovasc Imaging. 2018 Jan 1;19(1):39-46. doi: 10.1093/ehjci/jew321. PMID 28158582
- [Result] Gronlykke L, Ihlemann N, Ngo AT, Thyregod HG, Kjaergaard J, Korshin A, Gustafsson F, Hassager C, Nilsson JC, Sondergaard L, Ravn HB. Measures of right ventricular function after transcatheter versus surgical aortic valve replacement. Interact Cardiovasc Thorac Surg. 2017 Feb 1;24(2):181-187. doi: 10.1093/icvts/ivw350. PMID 27811168
- [Result] Jorgensen TH, Thyregod HG, Tarp JB, Svendsen JH, Sondergaard L. Temporal changes of new-onset atrial fibrillation in patients randomized to surgical or transcatheter aortic valve replacement. Int J Cardiol. 2017 May 1;234:16-21. doi: 10.1016/j.ijcard.2017.02.098. Epub 2017 Feb 24. PMID 28258844
- [Result] Thyregod HGH, Ihlemann N, Jorgensen TH, Nissen H, Kjeldsen BJ, Petursson P, Chang Y, Franzen OW, Engstrom T, Clemmensen P, Hansen PB, Andersen LW, Steinbruuchel DA, Olsen PS, Sondergaard L. Five-Year Clinical and Echocardiographic Outcomes From the NOTION Randomized Clinical Trial in Patients at Lower Surgical Risk. Circulation. 2019 Jun 11;139(24):2714-2723. doi: 10.1161/CIRCULATIONAHA.118.036606. Epub 2019 Feb 1. PMID 30704298
- [Result] Sondergaard L, Ihlemann N, Capodanno D, Jorgensen TH, Nissen H, Kjeldsen BJ, Chang Y, Steinbruchel DA, Olsen PS, Petronio AS, Thyregod HGH. Durability of Transcatheter and Surgical Bioprosthetic Aortic Valves in Patients at Lower Surgical Risk. J Am Coll Cardiol. 2019 Feb 12;73(5):546-553. doi: 10.1016/j.jacc.2018.10.083. PMID 30732707
- [Result] Geisler BP, Jorgensen TH, Thyregod HGH, Pietzsch JB, Sondergaard L. Cost-effectiveness of transcatheter versus surgical aortic valve replacement in patients at lower surgical risk: results from the NOTION trial. EuroIntervention. 2019 Dec 6;15(11):e959-e967. doi: 10.4244/EIJ-D-18-00847. PMID 31422922
- [Result] Jorgensen TH, Thyregod HGH, Ihlemann N, Nissen H, Petursson P, Kjeldsen BJ, Steinbruchel DA, Olsen PS, Sondergaard L. Eight-year outcomes for patients with aortic valve stenosis at low surgical risk randomized to transcatheter vs. surgical aortic valve replacement. Eur Heart J. 2021 Aug 7;42(30):2912-2919. doi: 10.1093/eurheartj/ehab375. PMID 34179981